CLINICAL TRIAL: NCT07304180
Title: Comparison of the Effects of Balance Exercises and Video Game-Based (Exergame) Exercises in Hemiplegia Rehabilitation
Brief Title: Exergame vs Balance Training in Hemiplegia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Ayşenur Çetinkaya, Lecturer (PhD), Halic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Acetinkaya008
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Hemiplegia; Exergaming; Exercise; Rehabilitation
MeSH Terms: conditions — Hemiplegia; Motor Activity | interventions — Exergaming

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1_Balance Exercise Group (Experimental): Participants in this group will receive conventional physiotherapy combined with balance exercise sessions twice a week for four weeks under the supervision of a physiotherapist.
  Interventions: Other: Balance exercise
- Group 2_Exergame Group (Experimental): Participants in this group will perform video-based exergame sessions in addition to conventional rehabilitation. The exergame intervention will be conducted using the Nintendo Switch Ring Fit Adventure game. Sessions will take place twice a week for four weeks under the supervision of a physiotherapist.
  Interventions: Other: Exergaming

INTERVENTIONS:
Other: Exergaming — Participants in this group will perform video-based exergame sessions in addition to conventional rehabilitation. These sessions will be conducted twice a week for four weeks, with each session lasting approximately 15-20 minutes under the supervision of a physiotherapist, using the Nintendo Switch Ring Fit Adventure game. The exergame program was designed by a specialist physiotherapist.
  Arms: Group 2_Exergame Group
Other: Balance exercise — Participants in this group will perform balance exercise sessions in addition to conventional rehabilitation. These sessions will be conducted twice a week for four weeks, with each session lasting approximately 15-20 minutes.
  Weeks 1-2: Weight shifting in parallel bars, marching in place within parallel bars, mini squats while holding the bars, tandem stance, and tandem and lateral walking in parallel bars.
  Week 3: Controlled weight shifting outside the parallel bars, tandem stance, marching in place, mini squats against a wall, backward walking in parallel bars, obstacle course walking, and kicking a stationary ball with the non-affected foot.
  Week 4: Picking up objects placed at different angles from a standing position, catching and throwing a ball, supported single-leg standing on the affected side, weight shifting on a balance board, kicking a moving ball with the non-affected foot, and obstacle walking tasks.
  Arms: Group 1_Balance Exercise Group

SUMMARY:
Hemiplegia rehabilitation is a long and demanding process, but with the right approach and patience, it is possible to regain lost functions and improve quality of life. Balance plays a critical role in helping stroke survivors regain independence. This randomized controlled study aims to compare the effects of balance exercises and video-based exergame training, in addition to conventional physiotherapy, on lower extremity functionality, balance, gait, daily living activities, quality of life, and fear of falling in patients with hemiplegia following stroke.

A minimum of 30 eligible participants will be randomly assigned to two groups:

Group 1 (Balance Exercise Group): Conventional physiotherapy plus balance exercises.

Group 2 (Exergame Group): Conventional physiotherapy plus video-based exergame sessions using the Nintendo Switch Ring Fit Adventure.

Both interventions will be conducted twice a week for four weeks under the supervision of a physiotherapist. Assessments will be performed before and after the intervention using standardized scales.

DETAILED DESCRIPTION:
Hemiplegia rehabilitation is not only a process of regaining lost motor functions but also a journey toward restoring independence and self-confidence. Balance improvement is one of the key components of this process, as it directly influences gait, mobility, and daily life participation. With technological advancements, exergame-based interventions have emerged as engaging and motivating tools that can complement traditional rehabilitation programs.

This study aims to compare the effectiveness of balance exercise training and exergame-based exercise programs when added to conventional physiotherapy in stroke patients with hemiplegia. Participants who meet the inclusion criteria and provide informed consent will be randomly allocated into two groups (n ≥ 15 per group).

Group 1 (Balance Exercise Group): Participants will perform balance exercises twice a week for four weeks, in addition to their conventional physiotherapy program, under the supervision of a physiotherapist.

Group 2 (Exergame Group): Participants will perform exergame sessions using Nintendo Switch Ring Fit Adventure twice a week for four weeks, alongside the same conventional physiotherapy program.

Outcome measures:

Lower extremity motor function: Fugl-Meyer Assessment for Lower Extremity Balance: Berg Balance Scale Functional mobility and gait: Functional Reach Test, Timed Up and Go Test, 10-Meter Walk Test Activities of daily living: Modified Barthel Index Quality of life: Stroke Impact Scale Fear of falling: Falls Efficacy Scale-International Assessments will be conducted at baseline and after the four-week intervention. Data analysis will be performed using the Statistical Package for Social Sciences (SPSS). Continuous variables will be expressed as mean ± standard deviation, and categorical variables as frequency and percentage. Depending on the normality of data distribution, appropriate parametric or non-parametric tests will be applied, with the level of significance set at p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 25 and 70 years.
* Have experienced either hemorrhagic or ischemic stroke.
* At least six months have passed since the stroke event.
* Have a Modified Rankin Scale score of 2 or 3.
* Able to stand independently.
* Able to walk at least 10 meters independently or with an assistive device.
* Able to sit and stand up independently.
* Have a Brunnstrom stage of at least 4 in both upper and lower extremities.
* Have a Brunnstrom stage of at least 3 in the hand.
* Have a Mini-Mental State Examination score greater than 24.
* Willing to voluntarily participate in the study.

Exclusion Criteria:

* History of more than one stroke.
* Participation in another exercise or rehabilitation program.
* Body Mass Index greater than 29.9.
* Cognitive, visual, or auditory impairments that interfere with -communication.
* Presence of other neurological disorders such as multiple sclerosis, Parkinson's disease, or spinal cord injury.
* Vestibular system disorders affecting balance (e.g., vertigo, CANVAS syndrome).
* Severe contractures, joint complications affecting movement, recent fractures, arthritis, or use of medications that may impair physical function.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | Baseline and after 4 weeks
  To assess postural control and fall risk. The scale consists of 14 items scored from 0 to 4, with a total possible score of 56. Higher scores indicate better balance ability. Assessments will be performed at baseline and after 4 weeks of intervention. Type: Continuous (Score range: 0-56)
Functional Reach Test | Baseline and after 4 weeks
  To measure dynamic balance and the ability to maintain a stable base of support while reaching forward. The distance between the starting and ending hand positions is recorded in centimeters. Higher values indicate better balance and lower fall risk. Type: Continuous (Distance in cm)

SECONDARY OUTCOMES:
Fugl-Meyer Assessment for Lower Extremity | Baseline and after 4 weeks
  Evaluates motor function of the lower extremity, including reflex activity, movement within and outside synergies, and coordination/speed. The total score ranges from 0 to 34, with higher scores indicating better motor function.
Timed Up and Go Test | Baseline and after 4 weeks
  Assesses functional mobility and dynamic balance. The time (in seconds) it takes to stand up from a chair, walk 3 meters, turn around, walk back, and sit down is recorded. Shorter times indicate better mobility.
10-Meter Walk Test | Baseline and after 4 weeks
  Measures walking speed over a 10-meter distance. The average time (in seconds) of three trials is recorded. Faster times indicate better walking performance.
Modified Barthel Index | Baseline and after 4 weeks
  Assesses independence in activities of daily living (e.g., feeding, dressing, mobility, toileting). Scores range from 0 to 100, with higher scores indicating greater independence.
Stroke Impact Scale | Baseline and after 4 weeks
  Evaluates quality of life after stroke across domains such as strength, hand function, mobility, daily activities, emotion, communication, participation, and memory. Scores range from 0 to 100, with higher values reflecting better perceived health status.
Falls Efficacy Scale-International | Baseline and after 4 weeks
  Assesses fear of falling during daily activities. The 16-item questionnaire is scored from 16 to 64, with higher scores indicating greater fear of falling.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur Çetinkaya, Principal Investigator — Halic University
Locations (1):
- Halic University, Istanbul, Eyupsultan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No